CLINICAL TRIAL: NCT04635969
Title: Determining the Effectiveness of Sexual Health and Development Education for Children With Intellectual Disability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aylin KURT (Other)
Responsible Party: Sponsor-Investigator, Aylin KURT, Research Assistant, Bulent Ecevit University
Organization: Bulent Ecevit University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2020/20
Record Dates: First submitted 2020-11-16; First posted 2020-11-19 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Child Behavior Problem; Intellectual Disability; Sexuality
MeSH Terms: conditions — Intellectual Disability; Sexuality | interventions — Sexual Health

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Children training (Experimental): All registered participants in intervention group will participate in a series of trainings on sexuality education.
  Interventions: Behavioral: Sexual Health and Development Education for Children With Intellectual Disability
- Control: No intervention (No Intervention): All registered participants in control group will not participate in a series of trainings on sexuality education.

INTERVENTIONS:
Behavioral: Sexual Health and Development Education for Children With Intellectual Disability — Sexual Health and Development Education for Children With Intellectual Disability: It is aimed to eliminate the problems related to personal care and cleaning of children with mental retardation, to learn the symptoms of adolescence and to learn the methods of protection from abuse.
  Arms: Experimental: Children training

SUMMARY:
By integrating sexuality and disability literatures, theories, and research, this study aims to: determine the effectiveness of sexual health and development education for children (12-18 years) with mild to moderate intellectual disability.

The research hypotheses are as follows:

H0: There is no significant difference between the intervention group and the control group in the mean score of the "Sexual Development Characteristics Scale of Children with Mentally Retardation in Adolescence" after the sexual health and development trainings given to children with intellectual disabilities.

H1: After the sexual health and development trainings given to children with intellectual disabilities, the mean score of the "Sexual Development Characteristics Scale of Children with Intellectual Disability in Adolescence" is significantly higher in the intervention group compared to the control group.

DETAILED DESCRIPTION:
By integrating sexuality and disability literatures, theories, and research, this study aims to: determine the effectiveness of sexual health and development education for children (12-18 years) with mild to moderate intellectual disability. The number of children in the groups will be analyzed based on another study in which one of the scales to be used in the study. According to the calculations made in the G-Power 3.1 Demo package program, when the effect size is accepted as 0.8, it was seen that at least 24 cases in each group (total 48 children) would be sufficient for 80% power. These children will be selected from 48 children who got the least score from the "Sexual Development Characteristics of Adolescent Children with Intellectual Disability Scale". In this way, the criteria sampling method will be used. In this way, the criteria sampling method will be used. Anticipated duration is one year.

The inclusion criteria of the children in the study are as follows:

* Being between the ages of 12-18
* Having mild to moderate mental disability
* Parent's agreement to participate in research
* Lack of speech and vision impairment
* Completing all trainings and follow-ups during the research period

For intervention group:

Once enrolled and consent is documented, eligible subject's will participate in the study for approximately three months. Participants will be expected to attend 8 training sessions over a two months period, each are up to half hours in length. Follow-up will be made at the beginning of the training, right after the last training and one month after the last training after the questionnaire. Data analysis will begin once all trainings have been completed. Investigators anticipate completing the study, including primary analyses, within one year from the date recruitment begins.

For control group:

Once enrolled and consent is documented, eligible subject's will participate in the study for approximately three months. Children in the control group will not be educated.Follow-up will be made at the beginning of the training, right after the last training and one month after the last training after the questionnaire. Data analysis will begin once all trainings have been completed. Investigators anticipate completing the study, including primary analyses, within one year from the date recruitment begins. After the study is completed, training will be provided to children in the control group in a way that will not affect the data of the study.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 12-18
* Mild to moderate intellectual disability
* Parents agree to participate in research.
* Lack of speech and vision impairment
* Completing all trainings and follow-ups during the research period

Exclusion Criteria:

* Not being between the ages of 12-18
* Having several intellectual disability
* Parents not agree to participate in research.
* Having speech and vision impairment
* Not completing all trainings and follow-ups during the research period

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Change of the mean scores obtained by the children in the intervention group from the "Sexual Development Characteristics Scale of Children with Intellectual Disability in Adolescence" before and after the trainings | 12 months
  "Sexual Development Characteristics Scale of Children with Intellectual Disability in Adolescence" will be completed before trainings that gathers quantitative data that will address attitudes about the children sexual health and development. The survey will also be completed at the end of trainings and one month after the final training. The quantitative data will be used to measure a change in the children's attitudes, and behaviors before and after the proposed intervention. Data will be analyzed using Statistical Package for the Social Sciences package program.
Difference between the mean score of the "Sexual Development Characteristics Scale of Children with Intellectual Disability in Adolescence" between intervention and control groups | 12 months
  "Sexual Development Characteristics Scale of Children with Intellectual Disability in Adolescence" will be completed before trainings that gathers quantitative data that will address attitudes about the children sexual health and development. The survey will also be completed at the end of trainings and one month after the final training. The quantitative data will be used to measure a change in the children's attitudes, and behaviors before and after the proposed intervention. Measurements will be made without training the control group. At the end of the study, Difference between the mean score of the "Sexual Development Characteristics Scale of Children with Intellectual Disability in Adolescence" between intervention and control groups will be examined. Data will be analyzed using Statistical Package for the Social Sciences package program.

SECONDARY OUTCOMES:
Children achieve 70% success in questions about education after each training | 12 months
  In order for children to move on to the next training, they must obtain 70% success points from post-training questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Special Therapy Special Education and Rehabilitation Center, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 12 months

REFERENCES:
- See also: Sexual Education and Development in Children with Intellectual Disability: Mothers' Opinions — http://link.springer.com/article/10.1007/s11195-020-09638-z